CLINICAL TRIAL: NCT03241069
Title: Dynamic Variation of Impedance Cardiography (ICG) a Diagnostic Tool of Acute Heart Failure (AHF) in Emergency Department (ED) Patients Admitted for Acute Dyspnea
Brief Title: Dynamic Variation of Impedance Cardiography(DYVIC) as a Diagnostic Tool of Acute Heart Failure (AHF)
Acronym: DYVIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: DYVIC
Record Dates: First submitted 2013-09-07; First posted 2017-08-07 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2020-10

CONDITIONS: Acute Heart Failure
Keywords: bio-impedance; BIOPAC system; dyspnea; acute heart failure
MeSH Terms: conditions — Dyspnea | interventions — Sitting Position; Valsalva Maneuver

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- patients with acute dyspnea (Experimental): patients presenting to the emergency department with acute onset dyspnea are assessed for acute heart failure using the bio impedance technology (BIOPAC system) to measure the cardiac output in different clinical situations.
  FIRST: the cardiac output (CO) is measured at the reference position. Inbetween each step the patient was put in the reference position during 5 minutes.
  Interventions: Other: Reference position
- the sitting position (Experimental): the patient is put at the sitting position and we measure the cardiac output by BIOPAC system (patient is put to a 90 degree sitting position during 1 to 2 minutes then the CO is measured 5 minutes later)
  Interventions: Other: Reference position; Other: Valsalva maneuver; Other: a passive leg rising maneuver
- a passive leg rising maneuver (Experimental): we make a passive leg rising and we measure the cardiac output by BIOPAC system (45 degree passive leg rising was done for 1 to 2 minutes and CO was measured during the maneuver 5minutes later.)
  Interventions: Other: Reference position; Other: sitting position; Other: Valsalva maneuver
- Valsalva maneuver (Experimental): the patient was asked to perform the Valsalva maneuver and we measure the cardiac output by BIOPAC system(patients are asked to perform the Valsalva maneuver by executing a forced blow into a manometer for 30 seconds and the CO is calculated during this test.)
  Interventions: Other: Reference position; Other: sitting position; Other: a passive leg rising maneuver

INTERVENTIONS:
Other: Reference position — patient is put in a 30 degree supine position during 5 minutes
  Other Names: baseline position
Other: sitting position — patient is put to a 90 degree sitting position during 1 to 2 minutes then the CO is measured
  Arms: Valsalva maneuver; a passive leg rising maneuver
Other: Valsalva maneuver — patients are asked to perform the Valsalva maneuver by executing a forced blow into a manometer for 30 seconds and the CO is calculated during this test.
  Arms: a passive leg rising maneuver; the sitting position
Other: a passive leg rising maneuver — we make a passive leg rising and we measure the cardiac output by BIOPAC system (45 degree passive leg rising was done for 1 to 2 minutes and CO was measured during the maneuver.)
  Arms: Valsalva maneuver; the sitting position

SUMMARY:
Dynamic variations of bio-impedance measured cardiac output using non pharmacologic intervention (sitting position, passive leg rising and valsalva maneuver) could be used to detect acute heart failure in patients admitted to the ED for dyspnea.

DETAILED DESCRIPTION:
Acute heart failure (AHF) is a frequent condition in emergency basis and is responsible of a big number of admissions, complications, and deaths.

despite advances in diagnostic techniques, AHF diagnosis still difficult and cost not effective.

Measurement of cardiac output (CO) is used as a way to evaluate global cardiac function and changes in CO may be used to identify a change in the hemodynamic status of a patient.

the gold standard of measuring CO is thermodilution catheterization, however this is an invasive technique that poses a risk to the patient.

Impedance cardiography (ICG) is a noninvasive method for measuring CO. it is performed by applying small electrical current to the chest, and through electrodes placed on the neck and sides.

the pulsatile flow of blood causes fluctuations in the current, and the device calculates CO from the impedance waveform.

In practice, the investigators connect the device "BIOPAC" by using four electrodes which the investigators place on the base of the neck (posterior face) and on the base of the thorax (posterior face).

The ECG recording is taken simultaneously with two other electrodes placed at the right upper limb and left lower limb.

In addition to detecting the electric current and the ECG, heart sounds are recorded using a sensor that is placed at the mitral site.

The various curves are displayed simultaneously and stored for analysis. Subjects were first placed in the semi sitting position 30°, and after 5 minutes had cardiac output measurements performed. (CO1)

A second cardiac output measurement was performed after 5 min of seated position. (C02)

Patients were then placed in the initial position, and after an additional 5 minutes had cardiac output measurements performed. (CO1')

A third set of measurement was obtained during 45° passive leg raising at 1 to 2 minutes.(CO3)

Patients were then placed in the initial position, and after an additional 5 minutes had cardiac output measurements performed. (CO1'')

During a Valsalva maneuver the investigators took the fourth cardiac output measurement. (CO4)

Patients were then placed in the initial position, and after an additional 5 minutes had cardiac output measurements performed. (CO1''')

Dynamic variations on bio-impedance measured CO using non pharmacologic intervention (sitting position, passive leg rising and Valsalva maneuver) could be used to detect AHF in patients admitted to the ED for dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* 18 year old or above
* non traumatic acute dyspnea

Exclusion Criteria:

* age <18 years,
* cardio respiratory arrest,
* coma,
* shock,
* need for inotropic or vasoactive drugs,
* mechanical ventilation,
* severe and sustained rhythm disorders,
* severe mitral valve disease,
* severe pulmonary arterial hypertension
* renal insufficiency with creatinine>150 μmol/l.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cardiac output rate measured by ICG before and during maneuvers in acute dyspneic patients between the AHF and non AHF groups | 12 hours
  The diagnostic performance of each maneuver is evaluated by calculating the CO in ml/min by bio-impedance technique and compare the values between patients with and without AHF and between baseline.
  The diagnosis of AHF is based on clinical, biological (BNP levels), radiological (chest X-ray) and cardiac ultrasound data.

SECONDARY OUTCOMES:
In hospital death | up to 10 days
  survivor or ,ot

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Samir, Profesor, Principal Investigator — University hospital of Monastir
Locations (1):
- Emergency Department, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: official department website — http://www.urgencemonastir.com